CLINICAL TRIAL: NCT07358052
Title: Current Status of Cardiovascular Diseases in Chinese Overweight/ Obesity Population: An Epidemiological Study (COPE）
Acronym: COPE
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: DAS-8633; U1111-1325-5282 (Other: World Health Organization ( WHO ))
Record Dates: First submitted 2025-11-24; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Part 1: Using CCDRFS data from 2013, 2018, and 2023, we will examine trends in CVD and key risk factors (hypertension, dyslipidemia, hyperglycemia, CKD) among overweight/obese adults, comparing prevalence by sex, urban/rural residence, and age to assess the impact of overweight/obesity on cardiovascular health for public health planning.
  Interventions: Other: No treatment given
- Part 2: Using CCDRFS 2023 data, we will perform a cross-sectional analysis to identify CVD risk factors in overweight and obese Chinese adults. We will: (1) compare characteristics of overweight/obese individuals with and without CVD, and (2) compare CVD patients who are overweight/obese versus normal weight. Odds ratios will be estimated to assess associations between risk factors and CVD within the overweight/obese group and to compare these associations against the normal-weight group. Subgroup and sensitivity analyses will be conducted to examine heterogeneity and robustness.
  Interventions: Other: No treatment given
- Part 3: We will link CCDRFS baseline data from 2013 and 2018 to the 2023 mortality follow-up database to estimate all-cause and cardiovascular mortality, population attributable fractions (PAF), and years of life lost (YLL) associated with overweight/obesity using Cox proportional hazards models.
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — No treatment given

SUMMARY:
This study is testing how overweight and obesity affect cardiovascular disease (CVD) prevalence, risk factors, and mortality among Chinese adults using nationally representative CCDRFS (China Chronic Disease and Risk Factor Surveillance) data. The purpose of the study is to characterize trends and determinants of CVD in adults with overweight or obesity and to quantify the excess mortality and population burden attributable to overweight/obesity. Participants will not receive any study medicine as this is an observational analysis of existing survey and mortality data. The study does not involve a new investigational drug; it analyses health and outcome data collected in routine practice and national surveys. The study will last for the duration needed to analyse the CCDRFS datasets and linked mortality follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
* Male or female, age above or equal to 18 years at the time of signing informed consent.
* Permanent residents (residing in the survey counties/cities/districts for ≥6 months) from the 2013, 2018, and 2023 CCDRFS surveys; With complete information from physical examinations, blood biochemical tests, and questionnaires, including:
* Demographic information (age, sex, urban/rural classification, etc.);
* Height, weight, waist circumference, blood pressure;
* Blood biochemical indicators (fasting/2-hour postprandial blood glucose, glycated hemoglobin, lipid panel: high density lipoprotein cholesterol, low-density lipoprotein cholesterol, triglycerides, total cholesterol, serum creatinine, etc.);
* Routine urine indicators: urine protein (or urine microalbumin); self-reported prevalence of CVD and major chronic diseases (e.g., hypertension, diabetes, dyslipidemia, etc.);
* Major behavioral risk factors (smoking, alcohol consumption, physical activity, dietary patterns, etc.);
* Information on concomitant medication use.

Exclusion Criteria:

- Exclusion criteria include missing core baseline or follow-up data relevant to each part. The medical conditions under investigation include overweight and obesity, along with their comorbidity with CVD and associated risk factors.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The subjects in this study are permanent residents aged 18 years and older who participated in the CCDRFS in 2013, 2018, and 2023. Eligible participants were permanent residents (residing ≥6 months) of the survey sites, which included 298 counties/districts across all 31 provinces, autonomous regions, and municipalities of mainland China.
Sampling Method: Non-Probability Sample
Enrollment: 551931 (Actual)
Dates: Start 2025-12-08 (Actual); Primary Completion 2025-12-12 (Actual); Study Completion 2025-12-12 (Actual)

PRIMARY OUTCOMES:
Primary End point | 2013-2023
  Primary outcome: prevalence of cardiovascular disease (CVD), defined as the proportion of participants reporting a physician diagnosis or self-reported history of coronary heart disease, stroke, heart failure, or peripheral artery disease. We will summarize how common CVD and related conditions are in the study population. Categorical variables (e.g., overweight/obesity, central obesity, prior diagnoses) will be reported as counts and percentages. Continuous variables (e.g., BMI, waist circumference) will be reported as n, mean, and SD. For each survey year (2013, 2018, 2023) we will compute crude and age-standardized, population-weighted prevalence estimates. Trends over time will be assessed using Joinpoint regression to estimate the Average Annual Percent Change (AAPC) with 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (2):
- China (2):
  - National Center for Chronic and Noncommunicable Disease Control and Prevention, Chinese CDC, Beijing, Beijing Municipality
  - Novonordisk Facility, Beijing

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com